CLINICAL TRIAL: NCT03555474
Title: Efficacy of the Theta Burst Stimulation and Functional Electrical Stimulation as Compared to Conventional Physiotherapy in Stroke Rehabilitation: A Randomized Controlled Trial
Brief Title: Efficacy of the Theta Burst Stimulation and Functional Electrical Stimulation in Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sree Chitra Tirunal Institute for Medical Sciences & Technology (Other Government)
Responsible Party: Principal Investigator, Dr. Chaturbhuj Rathore, Associate Professor, Sree Chitra Tirunal Institute for Medical Sciences & Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR/SO/HS/0032/2010
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Strokes Thrombotic
MeSH Terms: conditions — Thrombotic Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Single blind randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor was blinded to the type of intervention.

ARMS (3):
- Theta burst stimulation & Physiotherapy (Experimental): Patients were given theta burst stimulation (intermittent TBS (iTBS) to the affected hemisphere and continuous TBS (cTBS) to the unaffected hemisphere) along with physiotherapy. TBS was delivered for 3 times in a week for 4 weeks.The stimulation was given with an intensity of 60% of RMT. The iTBS protocol of 10 bursts of high-frequency stimulation (3 pulses at 50 Hz) was applied at 5 Hz every 10 second for a total of 600 pulses.
  Continuous TBS (inhibitory) was delivered to the unaffected hemisphere at the "hot-spot" with an intensity of 60% of RMT, 3 pulses at 50 Hz, repeated every 200 ms for a total of 600 pluses.
  Interventions: Procedure: Theta burst stimulation; Procedure: Physiotherapy
- Functional stimulation & Physiotherapy (Experimental): Patients in the functional electrical stimulation (FES) group received the electrical stimulation with electrodes positioned according to pattern 3 [Grasp/Flexion/Extension, PATT (pattern movement)] of the FES (F) mode of the instrument. The electrodes were connected to a stimulator controller unit that delivers alternating current at a frequency of 35 Hz and a pulse width of 200 µs, intensity 10~50 mA.
  The FES group stimulation session was given for 30 minutes for each day 3 times in a week (alternate days) for 4 weeks and it was concurrently synchronized with the physiotherapy.
  Interventions: Procedure: Functional Electrical Stimulation; Procedure: Physiotherapy
- Physiotherapy (Active Comparator): The following different physiotherapy regimens were followed for all the patients in the study.
  Passive/Active Range of Motion (ROM); Weight bearing and supportive reaction; Reaching activities; Grasping, holding and release; Upper extremity activities of daily living (ADL). Physiotherapy intervention was given to all the patients 5 days per week for 1 month. In addition, all patients continued to receive in-home physiotherapy 1 to 2 times per week by a home physiotherapist who was guided by the research physiotherapist.
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Theta burst stimulation — Patients were given intermittent TBS to the affected hemisphere and continuous TBS to the unaffected hemisphere for 4 weeks along with physiotherapy.
  Other Names: TBS
  Arms: Theta burst stimulation & Physiotherapy
Procedure: Functional Electrical Stimulation — Patients were given functional electrical stimulation of affected upper extremity for four weeks along with physiotherapy.
  Other Names: FES
  Arms: Functional stimulation & Physiotherapy
Procedure: Physiotherapy — Patients received active and passive physiotherapy of the affected extremity for four weeks.
  Other Names: PT

SUMMARY:
Approximately 50% of patients have persistent motor disability following stroke. Current treatment approaches with conventional physiotherapy have limited efficacy. Repetitive transcranial magnetic stimulation (rTMS) and Functional electrical stimulation (FES) have been shown to improve the neuronal plasticity and motor control in few preliminary studies. Their efficacy in human stroke subjects is unproven. We planned to study their efficacy in improving the motor functions of stroke patients in a randomized trial. Sixty consecutive haemodynamically stable adult patients with first ischemic stroke within last 7-30 days were randomized into three treatment groups to receive either physiotherapy alone, or physiotherapy combined with either FES or rTMS. Outcome was assessed using Fugl Meyer assessment for physical performance of upper limb. Three groups were compared for the outcome measures using intention to treat analysis.

DETAILED DESCRIPTION:
Background

Present management strategies involving conventional physiotherapy (PT) have limited efficacy in facilitating the motor recovery following stroke. Finding an effective intervention to improve motor recovery in individuals with hemiplegia is very important for improving the functional outcome and enabling independent living.

Following an injury, the brain undergoes significant reorganization of its functions resulting in functional recovery, which occurs over a period of weeks to months. This postlesional reorganization occurs mostly in the premotor cortex, dorsolateral prefrontal cortex and supplementary motor area which are thought to play the most important role in recovery following any type of brain injury. Treatment approaches which can facilitate this reorganization process by enhancing the cortical plasticity might have a very important role in improving the functional outcome following neuronal injury.

Both central and peripheral stimulation has potential to improve the cortical reorganization and functional recovery following acute stroke. Previous studies have established that following an acute stroke, the depressed excitability of the ipsilesional hemisphere can be increased by stimulating the ipsilesional hemisphere or by inhibiting the contralesional hemisphere.This happens because of the fact that one hemisphere has inhibitory effect on the other hemisphere through transcallosal inhibition. In preliminary studies, application of high frequency repetitive transcranial magnetic stimulation (rTMS) to motor cortex has been shown to produce an increase in corticospinal excitability leading to enhancement of motor functions. Theta Burst Stimulation (TBS), which is a novel method of delivering rTMS at lower intensities without the risk of any major adverse effects, has been found to be safe in chronic and acute stroke patients. In this regard, intermittent TBS (iTBS) has a stimulatory effect on the brain and continuous TBS (cTBS) has inhibitory effect on the brain. In preliminary studies, intermittent TBS (iTBS) applied to the ipsilesional hemisphere and continuous TBS (cTBS) applied to the contralesional hemisphere have been shown to improve the motor functions and corticospinal output in the paretic hands during experimental settings. However, long term effects of this strategy on functional outcome have not been previously studied. Similarly, functional electrical stimulation (FES), a form of peripheral stimulation, when applied to the paretic upper limb muscles has been shown to improve the upper limb functional activity in patients with acute or subacute stroke.

Thus both the TBS and FES has a potential of improving the motor functions and the functional outcome following ischemic stroke. However, these strategies have not been used in clinical setting and their usefulness in promoting motor recovery over and above that of conventional PT has not been proven. If proven to be useful, these techniques have a potential of improving the otherwise dismal functional outcome following stroke. The purpose of this study is to determine efficacy of TBS or FES as an adjunctive to physical therapy for the rehabilitation of stroke patients.

METHODS Study Setting and Participants This study is a single blind randomized controlled trial to assess the efficacy of TBS and FES in improving motor functions over and above that of standard PT following acute stroke. This study was carried out at the Department of Neurology, Sree Chitra Tirunal Institute for Medical Sciences and Technology, Trivandrum, Kerala, India. We recruited consecutive patients over a 28 months period from the outpatient clinics and inpatient wards. Patients with first ever ischemic stroke in middle cerebral artery territory who presented within 10 days to 30 days of onset and had ability to give informed consent and comprehend instructions were included in this study. All the patients underwent 1.5 T MRI and had documented single infarct in MCA territory with no other lesion. All the patients received standard medical and rehabilitative care including passive and active PT. The study was approved by the institutional ethics committee (SCT/IEC/223). All the patients provided written informed consent to undergo the trial. Consecutive patients who fulfilled the inclusion and exclusion criteria were randomized to one of the three groups: (1) those who received TBS as per the predefined protocol along with standard PT (Group A); (2) those who received FES as per the predefined protocol along with standard PT (Group B); and (3) those who received PT (PT) alone (Group C).

Random allocation and sequence generation The patients were randomly allocated into three groups by block randomization method. Concealed allocation was done by principle investigator who blindly allocated the subjects into different groups according to the block randomization table to receive the designated intervention

Blinding After providing the informed consent, a subject fulfilling the inclusion and exclusion criteria was initially assessed by first co-investigator for all the outcome measures and neurophysiological parameters. Patients who were eligible for the study were allocated to different intervention groups by principle investigator. Interventions were done by second co-investigator for all the subjects. Follow-up assessments were done by the first co-investigator who was blinded to the allocation to intervention groups.

Outcome measures As we mainly wanted to assess upper extremity functions, we used Fugl Meyer Assessment (FMA) scale as the primary outcome measure to assess the upper limb motor functions. This is a 66-point scale to evaluate upper limb functions, a standard tool for this purpose. In addition, we used Modified Rankin Scale (mRS) to assess global outcome, National Institute of Health Stroke Scale (NIHSS) to assess stroke severity and Barthel Index (BI) to assess activities of daily living. These three scales were used as secondary outcome measures.

Outcome scales were applied at baseline (T1) and then subsequent assessments were done at one month (T2), three months (T3), six months (T4) and at one year (T5) after the enrollment.

Sample size calculation Primary outcome measure for this study was the Fugl Meyer Assessment of upper limb functions at one year. Previous studies have shown that FMA score increases by 16.5 ± 9.4 at one year in control subjects.21 We hypothesized that for a clinically meaningful outcome, the intervention should produce an increase of 10 points over and above the control group. To achieve this, a sample size of 14 patients in each arm was required for a power of 80% with alpha fixed at 5%. In a previous study conducted at our institute, the post stroke mortality was 27.2 % at one year, of these 72.1% died within 10 days after the stroke.2 As have planned to include patients between 10 to 30 days of stoke onset, to account for the mortality rate of 7.6% after 10 days, the required sample size was 16 in each group. Considering a dropout rate of 20 %, we calculated a sample size of 20 patients in each group as adequate.

TMS Protocol We assessed resting motor threshold (RMT) for both the hemispheres at baseline using Magstim Rapid2 (Whitland, Wales, UK) stimulator with a figure-of-eight coil having an external loop diameter of 9 cm. After making the patient seated comfortably in an armchair, posterior-anterior orientation was used over the motor cortex (M1) to assume the optimal scalp position to elicit MEP in the contralateral first dorsal interosseous (FDI) muscle. RMT was assessed from ipsilesional hemisphere initially and followed by contralesional hemisphere as per the standard techniques. Surface electromyograms (EMGs) were recorded from the FDI muscles bilaterally using Ag-AgCl electrodes with a gain of 1-2 mv. Signals were filtered (10Hz-10 KHz), and then stored for off-line analysis. Audio-visual feedback of the EMG signal at high gain were given to assist subjects to maintain complete relaxation.

Patients in group A were subjected to TBS in addition to standard PT as described below. Intermittent TBS (iTBS), which is facilitatory, was given to the ipsilesional hemisphere and continuous TBS (cTBS), which is inhibitory, was given to contralesional hemisphere. The stimulation was given at an intensity of 60% of RMT. The iTBS protocol of 10 bursts of high-frequency stimulation (3 pulses at 50 Hz) was applied at 5 Hz every 10 s for a total of 600 pulses. When no MEP was elicited from the ipsilesional motor area (<0.05mV), 100% stimulator intensity as that of contralesional hemisphere was applied at the mirror location of the contralesional motor area.14 Continuous TBS was given with an intensity of 60% of RMT, 3 pulses at 50 Hz, repeated every 200 ms for a total of 600 pluses. Both iTBS and cTBS were delivered for three times in a week for four weeks.

Functional Electrical Stimulation. Electrical stimulation was given with Mega XP (Cybermedic Corporation, South korea). The patient received the electrical stimulation in sitting position with affected arm positioned over the pillow and electrodes were positioned according to pattern 3 [Grasp/Flexion/Extension, PATT (pattern movement)] of the FES (F) mode of the instrument. The stimulator controller unit of the machine could deliver alternating current at a frequency of 35 Hz, pulse width of 200 µs and intensity of 10~50 mA. The stimulator was set to deliver interrupted trains of pulses with the contraction and relaxation so as to simulate the lifting of upper limb in a functional position. The FES group stimulation session was given for 30 minutes for each day, 3 times in a week (alternate days) for 4 weeks and it was concurrently synchronized with the physical therapy.

Physical therapy treatment protocol The following physical therapy regimens were followed for all the patients in the study: Passive/Active Range of Motion (ROM) at all joints; weight bearing and supportive reaction; reaching activities; grasping, holding and release; and upper extremity activities of daily living (ADL). Physical therapy intervention was given to all the patients five days per week for one month. Modifications in the physical therapy was made by second co-investigator for each patient so that he or she was able to practice independently or with assistance from a family member after the intervention and was instructed to practice one hour per day. In addition, all patients continued to receive in-home physical therapy 1-2 times per week by a home care physical therapist who was guided by second co-investigator. The investigators used a logbook to monitor the actual amount of time that each patient exercised at home.

Statistical Methods We used descriptive statistics to summarize the data. Baseline comparability of groups, in terms of demographic data and baseline measurements were assessed with chi-square test and ANOVA. Non-normal data was subjected to reciprocal, logarithmic and exponential transformation and Komogrov-Smirnov and Shapiro-Wilks tests were done to assess normality. Parametric measures were analyzed with ANOVA followed by post-hoc analysis with bonferroni correction. Repeated measure ANOVA was used to find out between group and within group variability. Non parametric measures were analyzed with Kruskal Wallis test followed by post hoc analysis with Mann Whitney U test. Friedmans test and Kendalls W test was done to find the changes in three groups over a period of one year. All analyses were done using SPSS version 17.0 and p value of less than 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. First episode of ischemic stroke in the internal carotid artery territory defined on CT scan or MRI brain.
2. Presentation within 7 days to 1 month of stroke onset.
3. Age group between 18-70 years
4. Muscle power less than 3 according to Medical Research Council (MRC) Grading

Exclusion Criteria:

1. Brain stem stroke
2. Bilateral strokes
3. Hemorrhagic stroke
4. Significant joint deformity preventing effective physiotherapy
5. Severe internal carotid artery stenosis requiring intervention
6. Unstable cardiopulmonary status and other diseases which are likely to hamper the 1 year follow up
7. Patients with contraindication to transcranial magnetic stimulation
8. Patients with previous history of seizures
9. Patients on chronic anti-psychiatric and antidepressants drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10-05 (Actual); Primary Completion 2012-01-25 (Actual); Study Completion 2012-01-25 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment (FMA) scale | One year
  Fugl Meyer Assessment (FMA) scale, is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. We used upper limb motor function domain of FMA scale which is a 66 point domain with a score ranging from 0-66. The lower score indicates more severe disability in upper limb motor functions.

SECONDARY OUTCOMES:
Modified Rankin Scale | One year
  Modified Rankin Scale (MRS) is a 7 point (0-6) ranking scale to assess neurological disability. A score of 0 indicates normal functions with no symptoms while higher scores indicates more severe neurological disability.
National Institute of Health Stroke Scale (NIHSS) | One year
  National Institute of Health Stroke Scale (NIHSS) is used to assess severity of impairment caused by stroke. It consists of 11 items with each item having a score of 0-4, where 4 indicates more severe disability. The score from all items is summed up to achieve the final NIHSS score. The score ranges from 0-44 where higher score indicates more severe impairment.
Barthel Index | One year
  To assess activities of daily living

IPD SHARING:
Plan to Share IPD: Yes
Annonymized individual participant data will be shared on request. Pl. contact: cbrathore@gmail.com.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 3 months of request
Access Criteria: Data sharing request will be assessed by the investigator.